CLINICAL TRIAL: NCT05333562
Title: Effects of Motor Control Exercises With and Without Neural Mobilization on Postural Control of Older Adults
Brief Title: Motor Control Exercises and Neural Mobilization in Posture of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Raana Rubab
Record Dates: First submitted 2022-01-21; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Postural Control
Keywords: Motor control exercise; Neural mobilization; postural control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor control exercise (Other): Motor control exercise was given with total of 8 sessions for 30 min for 4 weeks twice a day. Each exercise was performed 10 repetitions for 10 sec.
  Interventions: Other: Motor control exercise
- Motor control exercise with neural mobilization (Active Comparator): this was given motor control exercise for 30 min, 4 weeks twice a day plus neural gliding applied for 3 sets of 10 repetitions on each session. Neural gliding applied 5 min before motor control exercise. Total 8 sessions were given
  Interventions: Other: Motor control exercise with mobilization

INTERVENTIONS:
Other: Motor control exercise — Motor control exercise was given with total of 8 sessions for 30 min for 4 weeks twice a day. Each exercise was performed 10 repetitions for 10 sec.
  Arms: Motor control exercise
Other: Motor control exercise with mobilization — this was given motor control exercise for 30 min, 4 weeks twice a day plus neural gliding applied for 3 sets of 10 repetitions on each session. Neural gliding applied 5 min before motor control exercise. Total 8 sessions were given
  Arms: Motor control exercise with neural mobilization

SUMMARY:
The aim of this research is to find and compare the effect of Motor control exercises with and without neural mobilization on postural control of older adults.

DETAILED DESCRIPTION:
Randomized controlled trials done at Bilqees Eidhi and Afiyat old age home Lahore.The sample size was 40. The subjects were divided in two groups, 20 subjects in Motor control exercise group and 20 in Motor control exercise with neural gliding group. Study duration was of 6 months. Sampling technique applied was purposive non probability sampling technique. Only 65-80 years of older adults included in study. Tools used in the study are time up and go test(TUG), Gait speed, Static balance and Quality of life(OPQOL35). Data was analyzed through SPSS 21.

ELIGIBILITY:
Inclusion Criteria

* Both male and female were included
* Older adults having age range from 60-80 years or older
* Adults whose score is more than 24 on mini mental state examination.
* Ambulate independently with or without a walking aid
* Adults who had permission from the institution's doctor to participate in exercise classes.

Exclusion Criteria:

* Patients with altered conscious level
* Adults who cannot ambulate (bed ridden patients)
* Patient with any neurological condition like stroke, multiple sclerosis and TBI
* Patients with severe orthopedic condition like fractures and rheumatoid arthritis
* Patient having any cardiac condition
* Adults walking with walking aids like sick and crutches
* Adults having vertigo or vestibular problems.
* Adults having history of recurrent falls.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Static balance test | first reading at 0 week
  Balance will be assessed using the Tandem stance (TS) test for static balance. The intraobserver reliability of the test is good with an ICC of 0.80.
Static balance test | final reading at end of 4 week
  Balance will be assessed using the Tandem stance (TS) test for static balance. The intraobserver reliability of the test is good with an ICC of 0.80.
Gait speed test | first reading at 0 week
  The 4-m gait speed test will use, and the beginning and the end of the test will mark on the floor. The intra-observer reliability of the gait speed test is excellent with an ICC of 0.91, a standard error of measurement of 0.06 m/s, and a minimum detectable difference (MDD) of 0.17 m/s.
Gait speed test | final reading at end of 4 week
  The 4-m gait speed test will use, and the beginning and the end of the test will mark on the floor. The intra-observer reliability of the gait speed test is excellent with an ICC of 0.91, a standard error of measurement of 0.06 m/s, and a minimum detectable difference (MDD) of 0.17 m/s.
Timed Up and Go test | first reading at 0 week
  Timing began when participants initiate standing and end when they sat down. The mean of the measurements will be use for statistical purposes. The inter-observer reliability is good with an ICC of 0.89, a standard error of measurement of 3.99 seconds, and an MDD of 11.06 seconds.
Timed Up and Go test | final reading at 4 week
  Timing began when participants initiate standing and end when they sat down. The mean of the measurements will be use for statistical purposes. The inter-observer reliability is good with an ICC of 0.89, a standard error of measurement of 3.99 seconds, and an MDD of 11.06 seconds.
Quality of life: (OPQOL 35) | first reading at 0 week
  OPQOL questionnaire, has been validated in a multiethnic community-dwelling older population in England. Cronbach's alpha coefficient for the Italian outpatient population enrolled in this study was found to be 0.78, i.e. above the 0.70 threshold of acceptability for internal consistency.
Quality of life: (OPQOL 35) | final reading at 4 week
  OPQOL questionnaire, has been validated in a multiethnic community-dwelling older population in England. Cronbach's alpha coefficient for the Italian outpatient population enrolled in this study was found to be 0.78, i.e. above the 0.70 threshold of acceptability for internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Binash Afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plaza-Manzano G, Cancela-Cilleruelo I, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL, Thoomes-de-Graaf M, Ortega-Santiago R. Effects of Adding a Neurodynamic Mobilization to Motor Control Training in Patients With Lumbar Radiculopathy Due to Disc Herniation: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2020 Feb;99(2):124-132. doi: 10.1097/PHM.0000000000001295. PMID 31464753
- [Background] Forrester LW, Roy A, Krywonis A, Kehs G, Krebs HI, Macko RF. Modular ankle robotics training in early subacute stroke: a randomized controlled pilot study. Neurorehabil Neural Repair. 2014 Sep;28(7):678-87. doi: 10.1177/1545968314521004. Epub 2014 Feb 10. PMID 24515923
- [Background] Aasa B, Berglund L, Michaelson P, Aasa U. Individualized low-load motor control exercises and education versus a high-load lifting exercise and education to improve activity, pain intensity, and physical performance in patients with low back pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2015 Feb;45(2):77-85, B1-4. doi: 10.2519/jospt.2015.5021. PMID 25641309
- [Background] Gurpinar B, Kara B, Idiman E. Effects of aquatic exercises on postural control and hand function in Multiple Sclerosis: Halliwick versus Aquatic Plyometric Exercises: a randomised trial. J Musculoskelet Neuronal Interact. 2020 Jun 1;20(2):249-255. PMID 32481240
- [Background] Silva-Batista C, Corcos DM, Kanegusuku H, Piemonte MEP, Gobbi LTB, de Lima-Pardini AC, de Mello MT, Forjaz CLM, Ugrinowitsch C. Balance and fear of falling in subjects with Parkinson's disease is improved after exercises with motor complexity. Gait Posture. 2018 Mar;61:90-97. doi: 10.1016/j.gaitpost.2017.12.027. Epub 2017 Dec 28. PMID 29310015
- [Background] Halliday MH, Pappas E, Hancock MJ, Clare HA, Pinto RZ, Robertson G, Ferreira PH. A randomized clinical trial comparing the McKenzie method and motor control exercises in people with chronic low back pain and a directional preference: 1-year follow-up. Physiotherapy. 2019 Dec;105(4):442-445. doi: 10.1016/j.physio.2018.12.004. Epub 2018 Dec 21. PMID 31204031
- [Background] Prasertsakul T, Kaimuk P, Chinjenpradit W, Limroongreungrat W, Charoensuk W. The effect of virtual reality-based balance training on motor learning and postural control in healthy adults: a randomized preliminary study. Biomed Eng Online. 2018 Sep 18;17(1):124. doi: 10.1186/s12938-018-0550-0. PMID 30227884
- [Background] Hamed A, Bohm S, Mersmann F, Arampatzis A. Exercises of dynamic stability under unstable conditions increase muscle strength and balance ability in the elderly. Scand J Med Sci Sports. 2018 Mar;28(3):961-971. doi: 10.1111/sms.13019. Epub 2018 Feb 6. PMID 29154407
- [Background] Stozek J, Rudzinska M, Pustulka-Piwnik U, Szczudlik A. The effect of the rehabilitation program on balance, gait, physical performance and trunk rotation in Parkinson's disease. Aging Clin Exp Res. 2016 Dec;28(6):1169-1177. doi: 10.1007/s40520-015-0506-1. Epub 2015 Dec 10. PMID 26661467
- [Background] Mateus A, Rebelo J, Silva AG. Effects of a Multimodal Exercise Program Plus Neural Gliding on Postural Control, Pain, and Flexibility of Institutionalized Older Adults: A Randomized, Parallel, and Double-Blind Study. J Geriatr Phys Ther. 2020 Jan/Mar;43(1):3-11. doi: 10.1519/JPT.0000000000000249. PMID 31569173